CLINICAL TRIAL: NCT01094171
Title: A Phase IV (Not Interventional), Open-label, Multicentre Study to Evaluate the Reactogenicity and Safety of Co-administration of GlaxoSmithKline Biologicals' DTPa (Infanrix) and IPV (Poliorix) Vaccines Administered as Three-dose Primary Immunisation Course at 3, 4.5 and 6 Months of Age in Healthy Children in Russian Federation
Brief Title: Study to Evaluate the Safety of Co-administration of GSK Biologicals' Poliorix and Infanrix in Healthy Children in Russia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113586; 2013-002804-15 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-26 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Poliomyelitis
Keywords: poliomyelitis; diphtheria; Primary immunization; pertussis; Children; tetanus
MeSH Terms: conditions — Poliomyelitis; Diphtheria; Whooping Cough; Tetanus

ARMS (1):
- Poliorix Group (Experimental): Subjects received 3 primary doses of PoliorixTM and InfanrixTM vaccines at 3, 4.5 and 6 months of age. All vaccines were administered intramuscularly in the anterolateral side of the left thigh (Poliorix) and the right thigh (Infanrix).
  Interventions: Biological: Poliorix TM; Biological: Infanrix TM

INTERVENTIONS:
Biological: Poliorix TM — Intramuscular administration, 3 doses
Biological: Infanrix TM — Intramuscular administration, 3 doses

SUMMARY:
The purpose of this study is to assess reactogenicity and safety of simultaneous administration of GSK Biologicals' inactivated poliomyelitis vaccine Poliorix and GSK Biologicals' DTPa-vaccine Infanrix vaccines in healthy children in Russian Federation in their first year of life according to National Calendar of Prophylactic Immunisation of Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 3 months including at the time of the vaccination.
* Written informed consent obtained from the parent of the subject.
* Healthy subjects as established by medical history and clinical examination and thermometry before entering into the study, that don't have contraindications for vaccination against diphtheria, tetanus, pertussis and poliomyelitis

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs from birth.
* Administration of immunoglobulins and/or any blood products from birth or planned administration during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the vaccination, except recombinant hepatitis B vaccine, Haemophilus influenzae type B vaccine and seasonal/pandemic influenza prophylactic.
* Participation in another clinical study at any time during the study, in which the subject has been or will be exposed to an investigational or a non-registered product (pharmaceutical product or device).
* Previous vaccination against diphtheria, tetanus, pertussis and poliomyelitis if by any reasons it was made in timeframe not stated by National Calendar of Prophylactic Vaccines of Russian Federation.
* Medical history of convulsions and progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Chronic diseases and serious congenital defects.
* Acute disease at the time of enrolment.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2010-12-03 (Actual); Primary Completion 2012-10-27 (Actual); Study Completion 2012-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Russia (2):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Yekaterinburg

REFERENCES:
- [Background] Romanenko VV et al. (2016) Safety and reactogenicity of inactivated vaccine for polio prevention (Poliorix ™) output and DTP vaccine (Infanrix ™) in a joint application for trehdozovoy scheme in healthy children in Russia. Ural Med Jq. 9(142):138-144.

RESULTS

PARTICIPANT FLOW:
Groups:
- Poliorix Group: Subjects received 3 primary doses of Poliorix™ and Infanrix™ vaccines at 3, 4.5 and 6 months of age. All vaccines were administered intramuscularly in the anterolateral side of the left thigh (Poliorix) and the right thigh (Infanrix).
Period: Overall Study
Arm/Group | Poliorix Group
Started | 400
Completed | 390
Not Completed | 10
Not completed — Lost to Follow-up | 2
Not completed — Informed consent withdrawal | 4
Not completed — Migration from the study area | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Poliorix Group
Number analyzed (Participants) | 400
Age, Continuous [Mean (Standard Deviation); unit: Months] | 3.40 (0.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 222

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any specified solicited local symptoms reported irrespective of intensity grade. Grade 3 pain was defined as considerable pain that prevented normal everyday activities. Grade 3 redness and swelling were defined as redness and swelling greater than (>) 20 millimeters (mm)
Time Frame: During the 4-day (Days 0 - 3) post vaccination period
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 400
Subjects
  [Any Pain] | 114
  [Grade 3 Pain] | 7
  [Any Redness] | 258
  [Grade 3 Redness] | 12
  [Any Swelling] | 152
  [Grade 3 Swelling] | 8

2. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed were Drowsiness, Irritability, Loss of appetite and Fever [Axillary temperature greater than or equal to (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any specified solicited general symptoms reported irrespective of intensity grade or relationship to vaccination. Any fever = oral temperature ≥ 37.5 degrees Celsius (°C). Grade 3 symptoms = symptoms that prevented normal activities. Grade 3 fever = oral temperature > 39.0°C.
Time Frame: During the 4-day (Days 0 - 3) post vaccination period
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 400
Subjects
  [Any Drowsiness] | 227
  [Grade 3 Drowsiness] | 15
  [Any Irritability] | 240
  [Grade 3 Irritability] | 20
  [Any Loss of appetite] | 133
  [Grade 3 Loss of appetite] | 10
  [Any Fever] | 69
  [Grade 3 Fever] | 1

3. Primary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0 - 30) post vaccination period
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 400
Subjects | 91

4. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed included medical occurrences that resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Month 4)
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 400
Subjects
  [Any SAEs] | 4
  [Related SAEs] | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Month 4; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 31-day (Days 0-30) post-vaccination period.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Poliorix Group
All-Cause Mortality (participants affected / at risk) | 0/400
Serious Adverse Events (participants affected / at risk) | 4/400
Other Adverse Events (participants affected / at risk) | 258/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poliorix Group (N=400)
Body temperature increased (General disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Periproctitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Poliorix Group (N=400)
Pain (General disorders) | 114
Redness (General disorders) | 258
Swelling (General disorders) | 152
Drowsiness (General disorders) | 227
Irritability (General disorders) | 240
Loss of appetite (General disorders) | 133
Fever (General disorders) | 69
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Body temperature increased (General disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.